CLINICAL TRIAL: NCT02428972
Title: Assessment of Cognitive Functions and Quality of Life in Patients Undergoing Surgery for Supratentorial Brain Tumor - a Comparison of Two Anaesthetic Techniques
Brief Title: Assessment of Cognitive Functions and Quality of Life in Patients Undergoing Surgery for Supratentorial Brain Tumor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Indu Kapoor, Doctor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IEC/NP-55/06.02.2015
Record Dates: First submitted 2015-04-08; First posted 2015-04-29 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Brain Tumor
Keywords: brain tumor; quality of life; cognition; anesthetic technique
MeSH Terms: conditions — Brain Neoplasms | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intravenous anesthesia (Experimental): propofol infusion @ 100-200 mcg/kg/min for maintenance of anesthesia
  Interventions: Drug: Propofol
- inhalational anesthesia (Active Comparator): sevoflurane MAC between 0.8-1.2 for maintenance of anesthesia
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — Propofol infusion @100-200 mcg/kg/min Fentanyl 1mcg/kg Vecuronium 0.1mg/kg Mannitol 1 gm/kg
  Other Names: 2,6-di(propan-2-yl)phenol
  Arms: intravenous anesthesia
Drug: Sevoflurane — MAC of Sevoflurane will be maintained between 0.8-1.2 Fentanyl 1mcg/kg Vecuronium 0.1mg/kg Mannitol 1 gm/kg
  Other Names: fluoromethyl hexafluoroisopropyl ether
  Arms: inhalational anesthesia

SUMMARY:
Primary brain tumors are highly associated with neurocognitive deficit and poor quality of life. There are number of studies indicating that brain tumors and their treatment modalities are often related to cognitive dysfunction. Apart from primary brain lesions, deficit can also occur because of Surgery, Radiotherapy, Chemotherapy, Antiepileptic and Corticosteroid treatment.Anaesthesia can also add to cognitive deficit in these patients. According to Ali et al. propofol provides better cognition scores compared to sevoflurane than isoflurane. The primary aim of their study was to compare the effects of 3 anesthetic regimens on hemodynamics and recovery characteristics of the patients. However in another study by Magni et al., the authors found that there is no difference in early cognitive function between sevoflurane and propofol. The aim of this prospective, randomized, open-label clinical trial was to compare clinical properties of sevoflurane-fentanyl with propofol-remifentanil anesthesia in patients undergoing supratentorial intracranial surgery. However both these studies evaluated the early cognitive function. The primary endpoint was to compare early postoperative recovery and cognitive functions within the two groups. They also evaluated hemodynamic events, vomiting, shivering, and pain. The literature is scarce on the severity, incidence and effect of anaesthetics on cognition and quality of life of these patients. Since most of the patients of brain tumor cannot be cured with surgery alone, improvement of quality of life and palliative care of the symptoms and cognitive function are important part of the treatment. Now the cognitive function has also been considered as an independent prognostic factor in the survival of patients of brain tumor. Cognitive function can also be related to tumor laterality. Patients with tumors in left hemisphere will have lower scores on verbal tests, whereas tumor in right hemisphere will have lower scores on facial recognition tests. Patients with tumors in the left hemisphere report more difficulty concentrating and those with right-hemisphere lesions,report more tension. Patients with primary brain tumors also experience serious challenges to their quality of life (QOL). These patients may face motor deficits, personality changes, cognitive deficits, aphasia, or visual field defects.

DETAILED DESCRIPTION:
Cognitive dysfunction is a common complication in primary or metastatic brain tumors and can be correlated to disease itself or various treatment modalities. The symptoms of cognitive deficits may include problems with memory, attention and information processing. There is a study which suggest that psychological distress is an important factor in reducing health related QOL in patients with brain tumors. However in some studies, depression was found to be another important independent predictor of QOL and has strong impact on survival. QOL is a extensive term that comprises physical or functional status, emotional well-being, and social well-being. It has been studied that QOL in patients with high-grade tumors do not differ those with grade III and grade IV tumors. Compared to patients with non-CNS cancers, brain tumor patients report more fatigue, cognitive dysfunction, and altered mood states. However, different levels of impairments have been observed in patients with brain tumors. To spread awareness of the illness, psychiatric interventions may be useful in these patients. Cognitive dysfunction may affect basic functions including attention or behavior or advanced functions like taking decisions or making plans. According to Yoshii Y et.al, Cognitive dysfunction before or after the surgery may not correlate with stage of tumor malignancy and degree of tumor resection. Cognitive function has been correlated to increased fatigue and depression in newly diagnosed malignant glioma patients.

After approval from Institute Ethics Committee and consent from the patient or guardian, we will include all adult patients between 18 - 65 years, of either gender scheduled for craniotomy for supratentorial brain tumors. We will exclude patients with a history of previous surgery for brain tumor, emergency surgery and non-consenting patients. To calculate the sample size we will first conduct a pilot study enrolling 30 patients, 15 in each group. Block randomization will be followed with blocks size of 10 patients. Patients will be randomized using the computer generated program. Demographic details will be noted. Patients will be adequately fasted prior to elective surgery. A standard anaesthesia protocol will be followed for all patients. Patients will be randomized in to two groups, Group S (Inhalational) and Group P (Intravenous). .Allocation of the group will be performed using an opaque sealed envelope method. General anaesthesia will be induced with Propofol 1.5 - 2 mg/kg.Anaesthesia will be maintained with either propofol (Group P) or Sevoflurane (Group S) along with mixture of oxygen and air [1:1] at flow rate of 2 liters per minute..The Minimum Alveolar Concentration (MAC) of Sevoflurane would be maintained between 0.8 - 1.2. In Group P, depth of anaesthesia will be guided by clinical signs such as tachycardia and hypertension. Intra-operative analgesia and muscle relaxation will be provided by boluses of fentanyl 1 mcg/kg and vecuronium 0.1 mg/kg, respectively. Intra-operative monitoring will include ECG, heart rate, invasive and non-invasive blood pressure, gases, end-tidal carbon dioxide, pulse oximetry, temperature and fluid input and output. Mannitol 1 gm/kg would be administered over a period of 20 minutes at the time of skin incision. Immediately after craniotomy, brain relaxation would be assessed using Brain Relaxation Score (BRS) in which the blinded surgeon will assess the condition of the brain as 1 = perfectly relaxed, 2 = satisfactorily relaxed, 3 = firm (leveled) brain, 4 = bulging brain.(27)At the end of surgery, propofol would be discontinued at the beginning of skin closure and Sevoflurane at the end of the skin closure. Neuromuscular block will be reversed with neostigmine 0.1 mg/kg and glycopyrrolate 0.01 mg/kg. If patients are planned for elective mechanical ventilation in the post-operative period, neuromuscular block will not be reversed.

Emergence and extubation times will be noted. Emergence time is defined as time from discontinuation of anaesthetic to time to follow verbal commands and eye opening. Extubation time is defined as time from anesthetic discontinuation to tracheal extubation. Recovery of the patient will be assessed using the modified Aldrete score. Intraoperative and postoperative complications, if any, will be noted. Various complications (tachycardia, bradycardia, hypotension, hypertension) will be treated with fentanyl, atropine, mephentramine and labetalol. All patients will be shifted to the ICU for supportive care and further management. Cognitive functions would be assessed preoperatively (baseline), between 2 to 3 hours postoperative, 24 hours post-operative, three months and six month. Quality of life (QOL) will be assessed at three month, six month and one year. Cognitive function will be assessed for memory, learning, executive functioning, sustained attention and verbal fluency and QOL by neuro-psychologist as shown in Appendix below. The difference of brain relaxation by two grades between the two study groups will be considered clinically significant and sample size calculated on this basis.

Appendix

NEUROPSYCHOLOGICAL ASSESSMENT

FUNCTION TEST [1]: Memory & Learning, TEST: Auditory Verbal Learning Test (AVLT), DOMAINS: Verbal Memory, Learning & Retention, TIME TAKEN: 20 minutes, AVAILABILITY: Property of Clinical Neuropsychology (CNP). FUNCTION TEST [2]: Executive Functioning, TEST: Stroop Test, DOMAINS: Response Inhibition, perceptual set, TIME TAKEN:10 minutes, AVAILABILITY: Property of Clinical Neuropsychology (CNP). FUNCTION TEST [3]: Speed, TEST: Digit Symbol Substitution Test (DSST), DOMAINS: Mental speed, visuomotor coordination, motor persistence, sustained attention, response speed, TIME TAKEN:10 minutes, AVAILABILITY: Property of Clinical Neuropsychology (CNP). FUNCTION TEST [4]: Verbal Fluency, TEST: Controlled Oral Word Association (COWA) Test, DOMAINS: Phonemic fluency, language, TIME TAKEN:5 minutes, AVAILABILITY: Property of Clinical Neuropsychology (CNP). FUNCTION TEST [5]: Quality of life, TEST: WHO QOL - BREF, DOMAINS: QOL, TIME TAKEN:5 minutes, AVAILABILITY: Property of Clinical Neuropsychology (CNP).

ELIGIBILITY:
Inclusion Criteria:

* All adult patients between 18 - 65 years, of either gender scheduled for craniotomy for supratentorial brain tumors.

Exclusion Criteria:

* Patients with a history of previous surgery for brain tumor, emergency surgery and non-consenting patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Cognitive functions | Six month.

SECONDARY OUTCOMES:
Adverse events | 24 hours
  Number of patients suffering delay in emergence, hemodynamic instability, nausea, vomiting, pneumocephalus.

CONTACTS AND LOCATIONS:
Overall Officials: Indu Kapoor, MD, Principal Investigator — All India Institute of Medical Sciences

IPD SHARING:
Plan to Share IPD: No